CLINICAL TRIAL: NCT04685473
Title: A Phase I Study of Safety, Tolerability and Pharmacokinetics of T-1101 (Tosylate) Capsules in Subjects With Advanced Refractory Solid Tumors
Brief Title: Safety and Tolerability Study for T-1101 (Tosylate) Capsules to Treat Advanced Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taivex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAI-003
Record Dates: First submitted 2020-12-13; First posted 2020-12-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Advanced Refractory Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T-1101 (Tosylate) (Experimental)
  Interventions: Drug: T-1101 (Tosylate)

INTERVENTIONS:
Drug: T-1101 (Tosylate) — T-1101 (Tosylate) Capsule

SUMMARY:
T-1101 (Tosylate) is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by Taivex Therapeutics Corp. T-1101 (Tosylate) is a potent anti-cancer agent in numerous human cancer cell lines. In addition, oral administration of T-1101 (Tosylate) showed tumor growth inhibition in different mouse xenograft models of human cancers. In this study, safety, tolerability and pharmacokinetic (PK) of T-1101 (Tosylate) capsules will be evaluated and also the recommended dose and regimen(s) to initiate Phase 2 will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed and dated informed consent form indicating that the subject has been informed of all pertinent aspects of the study
2. Histologically and cytologically confirmed advanced malignancies that are refractory to standard treatments
3. Solid tumors that are measurable or evaluable as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion) unless increase in size is observed following completion of radiation therapy
4. Have a life expectancy of ≥3 months in the investigator's opinion
5. Females or males ≥ 20 years old
6. ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
7. Recovered from prior treatment-related toxicity to at least grade 1 with exception of alopecia
8. Adequate organ function as defined by the following criteria:

   1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 3 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
   2. Total serum bilirubin ≤ 1.5 x ULN
   3. Absolute neutrophil count (ANC) ≥ 1500/μL
   4. Platelets ≥ 100,000/μL
   5. Hemoglobin ≤ 9.0 g/dL
   6. Creatinine clearance (CrCl) ≥ 50 mL/min CrCl = [(140 - age (year)) x weight (kg)] / (serum creatinine x 72) (x 0.85 for females)
9. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

1. Major surgery within 4 weeks prior to starting T-1101 (Tosylate).
2. Subjects received any of the following anti-cancer therapies:

   1. Anti-cancer radiation therapy within 2 weeks prior to starting T-1101 (Tosylate).
   2. Palliative radiation (≤ 10 fractions) within 48 hours prior to the screening
   3. Any systemic cytotoxic chemotherapy within 2 weeks or 5 half-lives (whichever is greater) prior to starting T-1101 (Tosylate)
   4. Any target therapy within 2 weeks prior to starting T-1101 (Tosylate)
3. Any interventional treatments in another clinical trial within 2 weeks or 5-half-lives (whichever is greater) prior to starting T-1101 (Tosylate)
4. Documented or suspected brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease
5. Any of the following within 6 months of starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack
6. Ongoing cardiac dysrhythmias of ≥ NCI CTCAE v5.0 grade 2, or atrial fibrillation of any grade
7. Hypertension that cannot be controlled by medications (> 160/100 mm-Hg despite optimal medical therapy).
8. Known human immunodeficiency virus (HIV) infection
9. A positive test for hepatitis B (HBsAg) or hepatitis C (anti-HCV (hepatitis C virus) antibody), unless the HBV (hepatitis B virus) DNA level and/or HCV RNA level is below the limit of detection.
10. Men and women of childbearing potential who are unwilling to use highly effective contraceptive methods during the study period.

    Highly effective contraceptive methods include implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, surgical sterilization or a partner who is sterile.
11. If females, patient is pregnant or breastfeeding
12. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgement of the investigator and/or sponsor, excess risk associated with study participation or study drug administration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of T-1101 (Tosylate) in Participants with Advanced Cancers Refractory to Standard Therapy | The first 28-day cycle
  MTD is highest dose level of 30% target toxicity rate and the MTD will be determined based on the occurrence of the dose-limiting toxicity (DLT) assessed using toxicity data during Cycle 1 (the first 28 days).
  When following toxicity events occur within the first 28-day cycle, these toxicity will be defined as DLT.
  1. Hematological toxicities : prolonged grade 4 neutropenia for >7 days, grade 3 febrile neutropenia (an ANC < 1000/mm3 with a single temperature of > 38.3°C or a sustained temperature of > 38°C for more than 1 hour), grade 4 febrile neutropenia (febrile neutropenia with life-threatening consequences; urgent intervention indicated), Grade 3 or 4 neutropenia with IV treatment for infection and grade 3 thrombocytopenia with bleeding or grade 4 lasting 7 days.
  2. Non-hematological toxicities: grade 3 or 4 toxicities, Nausea and vomiting or diarrhea must persist at grade 3 or 4 despite maximal medical therapy.

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) to the time of the last measurable concentration and to infinity of T-1101 (Tosylate) | Selected time points during first 28-day cycle
  Area under the plasma concentration versus time curve to the time of the last measurable concentration (AUC0-last) of T-1101 (Tosylate) will be estimated using non-compartmental analysis. If data permit, area under the plasma concentration versus time curve to infinity (AUC0-∞) will be also estimated.
Pharmacokinetics: Time to maximum plasma concentration (Tmax) and terminal half-life (T½) of T-1101 (Tosylate) | Selected time points during first 28-day cycle
  Time to maximum plasma concentration (Tmax) of T-1101 (Tosylate) will be estimated using non-compartmental analysis. If data permit, terminal elimination half-life (T½ ) will be also estimated.
Pharmacokinetics: Oral plasma clearance (CL/F) of T-1101 (Tosylate) | Selected time points during first 28-day cycle
  Oral plasma clearance (CL/F) of T-1101 (Tosylate) will be estimated using non-compartmental analysis.
Pharmacokinetics: Apparent volume of distribution (Vd/F) of T-1101 (Tosylate) | Selected time points during first 28-day cycle
  Apparent volume of distribution (Vd/F) of T-1101 (Tosylate) will be estimated using non-compartmental analysis.
Clinical Tumor Response of T-1101 (Tosylate) in Participants with Advanced Cancers | Up to 2 years
  Categorization of response based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: No